CLINICAL TRIAL: NCT01787097
Title: GR Activity in Induced Sputum Macrophages, and a Change in Inflammatory Biomarkers 2-hours After a Single Dose of Either Symbicort®/Budesonide/Formoterol or in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effect of Symbicort ® on GR in Sputum in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D589BC00004; 2010-020440-35 (EudraCT Number)
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Chronic Obstructive Lung Disease
Keywords: Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COPD (Active Comparator): Participants with COPD
  Interventions: Drug: Formoterol 24ug
- Symbicort® total dose 400ug/12ug (Active Comparator): Symbicort® total dose 400ug/12ug: is a combination of FORM (6ug) and ICS (Budesonide, (BUD) 200ug)
  Interventions: Drug: Symbicort® total dose 400ug/12ug
- Symbicort® total dose 800ug/24ug (Active Comparator): Symbicort® total dose 800ug/24ug: is a combination FORM (12ug) and BUD (400ug) at a higher-dose
  Interventions: Drug: Symbicort® total dose 800ug/24ug
- BUD total dose 800ug (Active Comparator): BUD total dose 800ug: is an intermediate dose of ICS
  Interventions: Drug: BUD total dose 800ug

INTERVENTIONS:
Drug: Symbicort® total dose 400ug/12ug — Symbicort® is combination of formoterol 400ug and budesonide 12ug. Single dose
  Arms: Symbicort® total dose 400ug/12ug
Drug: Symbicort® total dose 800ug/24ug — Symbicort® is combination of formoterol 800ug and budesonide 24ug. Single dose
  Arms: Symbicort® total dose 800ug/24ug
Drug: Formoterol 24ug — Turbuhaler
  Arms: COPD
Drug: BUD total dose 800ug — Turbuhaler
  Arms: BUD total dose 800ug

SUMMARY:
The purpose of the research (or "knowledge gap" this research is designed to fill) is to understand the science of how the combination therapy of 2 drugs (inhaled longacting beta-agonists(LABA) and inhaled corticosteroids (ICS), which are commonly used in chronic obstructive pulmonary disease (COPD) patients, is better than each drug alone. ICS and LABA both have antiinflammatory properties; that is, they dampen the inflammation in the cells of the airways in the lungs. The combination of LABA and ICS has also been shown to improve clinical effectiveness in asthma patients. The addition of a LABA to LOW doses of ICS has been shown to be more clinically beneficial in asthma than the use of HIGH doses of ICS alone. This has allowed a reduction in the total ICS dose and minimised the adverse side effects of inhaled corticosteroids. Recent evidence suggests that the use of combination therapy of LABA and ICS may also improve clinical effectiveness in COPD patients.

Investigators will address this hypothesis by examining the inflammation cells of COPD direct from the site of disease (the airways) by looking at sputum/mucus. This research will build on the existing knowledge of the science of how these drugs work in asthma and COPD and allows us to understand the molecular science, which may support new future drug targets for patients with COPD, which are greatly needed.

DETAILED DESCRIPTION:
Corticosteroids exert their effects by binding to a cytoplasmic glucocorticoid receptor (GR). The inactive GR is bound to a protein complex that includes heat shock protein hsp90, acting as molecular chaperones to prevent the nuclear localisation of unoccupied GR.

GR binding to the palindromic promotor induces the transcriptional induction of anti-inflammatory genes such as mitogen-activated protein kinase phosphatase-1 (MKP-1) and secretory leukocyte protease inhibitor (SLPI). GR-steroid complex also binds to negative GRE sequences, resulting in inhibition of pro-inflammatory mediators, such as IL-6. More importantly, GR binds transcription factor with recruitment of histone deacetylase (HDAC) and inhibits wide range of pro-inflammatory cytokines. By this process of transrepression, corticosteroids reduce such pro-inflammatory cytokines as tumour necrosis-alpha (TNF-alpha) and interleukin-8 (IL-8) in asthmatic patients whereas they are far less effective in chronic obstructive pulmonary disease (COPD) patients.

The combination of inhaled corticosteroids (ICS) and long acting beta 2-agonists (LABAs) has been shown to improve clinical effectiveness and anti-inflammatory properties in asthma. The addition of a LABA to low dose ICS has been shown to be more clinically beneficial in asthma than the use of high dose ICS, allowing a reduction in ICS dose and minimising and adverse side effects of corticosteroids. Recent evidence suggests that this may also be the case in COPD.

ICS such as budesonide, beclomethasone and fluticasone have been used in combination with LABA's such as formoterol and salmeterol. These combination treatments are established in national guidelines for treating patients with asthma and also, COPD. The combination of formoterol and budesonide (Symbicort ®, Astra Zeneca) will be studied in this project.

Evidence suggests that LABAs enhance GR function in vitro. In an asthmatics study, the combination of formoterol and budesonide (Symbicort ®, Astra Zeneca) was as effective as high dose ICS on GR activation, gene transactivation and transrepression. However, the precise mechanisms for this enhanced effectiveness are unknown, although priming of the steroid receptor (GR) by LABAs may be important.

Investigators have developed a novel method of measuring GR-GRE binding activity in sputum using an enzyme immunosorbent assay system. This method, together with the measurements of some functional readouts, will help us to understand some of the mechanisms of steroid and GR interactions using non-invasive methods of assessment of the airways. This may provide insight into the mechanisms of corticosteroid action and whether the addition of a LABA to ICS can alter molecular patterns, which may explain the observed beneficial action of combination therapy seen in patient studies in vivo. This may allow a scientific basis to explore future drug interactions that may be helpful in patients, particularly those patients whose disease tends to be severe and may be unresponsive to standard therapies for COPD and/or where high dose ICS have little beneficial clinical effect and have led to side-effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (n=30) with chronic obstructive pulmonary disease (COPD) with mild-to-moderate disease severity (GOLD 1 and 2 guidelines). The post-bronchodilator FEV1 will be used in the criteria to define GOLD severity (reference 7/Table 1).
2. Aged 38-80 years inclusive
3. FEV1 <15% reversibility (not % predicted) and/or an increase of <200 ml after inhaled β2-agonists (400 μg salbutamol)
4. Patients will be allowed to use their current short-acting β2-agonists (SABA) and long-acting β2-agonists (LABA) and short-acting muscarinic-antagonist (SAMA) and long-acting muscarinic-antagonists (LAMA). However they should refrain from short-acting β2-agonists (SABA) and short-acting muscarinic-antagonist (SAMA) for 6 hours before the study visit and for long-acting β2-agonists (LABA) and long-acting muscarinic-antagonists (LAMA) at least 12 hours before the study visit, unless needed by the patient's clinical condition.
5. Theophylline (an oral tablet bronchodilator) will be required to be stopped at least 3 days prior to start of Study Visit one, and patients will not be allowed this treatment during the study as it may affect the GR response and the bronchodilator (lung function, spirometry) responses.
6. Capable of giving informed consent.

Exclusion Criteria:

1. As a result of the medical interview, physical examination or screening investigations, the Physician Responsible considers the volunteer unfit for the study.
2. Patients who have a clinical diagnosis of Asthma, as decided by the Study Investigators, as this does not fulfil the diagnosis of chronic obstructive pulmonary disease (COPD).
3. Patients who have had a history of an upper or lower respiratory infection (including sinusitis) within 4 weeks prior to study entry, as this can affect the breathing response.
4. Patients who have received oral or parenteral steroids within 4 weeks prior to study entry, as this can affect the breathing response and signifies that their condition needs to be controlled better.
5. Patients who have been hospitalised for a COPD exacerbation within 1 month of study entry and/or has received antibiotics within 4 weeks of study entry, as this signifies that their condition needs to be controlled better.
6. Patients taking any regular medication that is contraindicated (as indicated in the British National Formulary) in those about to receive the study medications listed in this protocol; other than the oral contraceptive pill.
7. Any evidence of a positive pregnancy urine test for female volunteers or females who are pregnant or lactating or are likely to become pregnant during the trial. Women of child-bearing potential may be included in the study if, in the opinion of the investigator, they are taking adequate contraceptive precautions (which will be directly enquired at the screening visit).
8. Patients who have a history of drug allergy which, in the opinion of the Unit Physician, contraindicates his/her participation in the study.
9. Patients with a known or suspected allergy to corticosteroids or any component of the formulations and/or suspected hypersensitivity to inhaled corticosteroid (this will be asked directly at the screening visit).
10. Patients who regularly, or on average, drink more than 21 units of alcohol (males) and 14 units of alcohol (female) per week (this will be asked directly at the screening visit).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar S Usmani, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton and Harefield NHS trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ito K, Barnes PJ, Adcock IM. Glucocorticoid receptor recruitment of histone deacetylase 2 inhibits interleukin-1beta-induced histone H4 acetylation on lysines 8 and 12. Mol Cell Biol. 2000 Sep;20(18):6891-903. doi: 10.1128/MCB.20.18.6891-6903.2000. PMID 10958685
- [Background] Keatings VM, Jatakanon A, Worsdell YM, Barnes PJ. Effects of inhaled and oral glucocorticoids on inflammatory indices in asthma and COPD. Am J Respir Crit Care Med. 1997 Feb;155(2):542-8. doi: 10.1164/ajrccm.155.2.9032192.
- [Background] Culpitt SV, Maziak W, Loukidis S, Nightingale JA, Matthews JL, Barnes PJ. Effect of high dose inhaled steroid on cells, cytokines, and proteases in induced sputum in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1999 Nov;160(5 Pt 1):1635-9. doi: 10.1164/ajrccm.160.5.9811058. PMID 10556133
- [Background] Calverley P, Pauwels R, Vestbo J, Jones P, Pride N, Gulsvik A, Anderson J, Maden C; TRial of Inhaled STeroids ANd long-acting beta2 agonists study group. Combined salmeterol and fluticasone in the treatment of chronic obstructive pulmonary disease: a randomised controlled trial. Lancet. 2003 Feb 8;361(9356):449-56. doi: 10.1016/S0140-6736(03)12459-2. PMID 12583942
- [Background] Calverley PM, Boonsawat W, Cseke Z, Zhong N, Peterson S, Olsson H. Maintenance therapy with budesonide and formoterol in chronic obstructive pulmonary disease. Eur Respir J. 2003 Dec;22(6):912-9. doi: 10.1183/09031936.03.00027003. PMID 14680078
- [Background] Essilfie-Quaye S, Ito K, Ito M, Kharitonov SA, Barnes PJ. Comparison of Symbicort(R) versus Pulmicort(R) on steroid pharmacodynamic markers in asthma patients. Respir Med. 2011 Dec;105(12):1784-9. doi: 10.1016/j.rmed.2011.08.020. Epub 2011 Sep 7. PMID 21903370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was enrolled January 2013. 4 participants withdrew before randomisation.
Groups:
- Formoterol 24ug: The first intervention is Formoterol (FORM) total dose 24ug, then Symbicort® total dose 400ug/12ug, then Symbicort® total dose 800ug/24ug, then BUD total dose 800ug
- Symbicort® Total Dose 400ug/12ug: The first intervention is Symbicort® total dose 400ug/12ug, then Formoterol (FORM) total dose 24ug, then Symbicort® total dose 800ug/24ug, then BUD total dose 800ug
- Symbicort® Total Dose 800ug/24ug: The first intervention is Symbicort® total dose 800ug/24ug, then Formoterol (FORM) total dose 24ug, then Symbicort® total dose 400ug/12ug, then BUD total dose 800ug
- BUD Total Dose 800ug: The first intervention is BUD total dose 800ug, then Symbicort® total dose 800ug/24ug, then Formoterol (FORM) total dose 24ug, then Symbicort® total dose 400ug/12ug
Period: Overall Study
Arm/Group | Formoterol 24ug | Symbicort® Total Dose 400ug/12ug | Symbicort® Total Dose 800ug/24ug | BUD Total Dose 800ug
Started | 8 (Study started in 2012/2013) | 7 | 7 | 9
Completed | 7 (Study completed) | 7 | 7 | 9
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Symbicort®, Formoterol, Budesonide: All Patients will receive randomly one-off dose of the following treatments:
  1. Formoterol (FORM) total dose 24ug: is a LABA chosen at a higher clinical dose to determine whether this treatment can achieve an effective treatment response on GR in sputum cells compare to treatments 2 and 3.
  2. Symbicort® total dose 400ug/12ug: is a combination of FORM (6ug) and ICS (Budesonide, (BUD) 200ug) at a lower-dose to determine whether this combination can have an effect on GR in sputum cells compare to treatment 4, 1 and 3.
  3. Symbicort® total dose 800ug/24ug: is a combination FORM (12ug) and BUD (400ug) at a higher-dose, chosen to compare the effect on GR with treatment 4 and 1
  4. BUD total dose 800ug: is an intermediate dose of ICS chosen for comparison with treatments 2 and 3 on GR.
  Symbicort®, Formoterol, Budesonide: Formeterol is Long acting beta 2-agonist (LABA) whereas Budesonide is inhaled corticosteroids (ICS).
Arm/Group | Symbicort®, Formoterol, Budesonide
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30
Pre-bronchodilator FEV1 (% pred.) [Median (Inter-Quartile Range); unit: % pred.] | 62 [55 to 70]
Pre-bronchodilator FVC (% pred.) [Median (Inter-Quartile Range); unit: % pred.] | 93 [83 to 103]
Sputum CXCL8 [Median (Inter-Quartile Range); unit: ng/mL] | 2.3 [1.4 to 4.0]

OUTCOME MEASURES:

1. Primary Outcome: GR-GRE Binding (Relative to Baseline)
Description: Enzyme immunosorbent assay system
Time Frame: Screening visit and 2 hours post inhalation of treatment
Population: Low patient numbers due to the fact that only a small number of patients were able to produce sputum that was of sufficient quality to undertake analysis, furthermore, sputum production between patient visits was highly variable.
Measure: Mean (Standard Error); unit: Fold activation
Groups:
- Formoterol (FORM) Total Dose 24ug: Participants received Formoterol (FORM) total dose 24ug
- Symbicort® Total Dose 400ug/12ug: Participants received 2 puffs of a combination of formoterol (6ug) and ICS (Budesonide, (BUD) 200ug)
- Symbicort® Total Dose 800ug/24ug: Participants received 2 puffs of a combination of formoterol (12ug) and budesonide (400ug)
- Pulmicort 800ug: Participants received 2 puffs of Budesoinde 400g (total dose 800ug)
Arm/Group | Formoterol (FORM) Total Dose 24ug | Symbicort® Total Dose 400ug/12ug | Symbicort® Total Dose 800ug/24ug | Pulmicort 800ug
Number analyzed (Participants) | 5 | 6 | 6 | 7
Fold activation | 1.1 (0.1) | 1.8 (0.1) | 2.3 (0.4) | 2.1 (0.2)
Statistical Analysis 1: Comparison: Symbicort® Total Dose 400ug/12ug vs Symbicort® Total Dose 800ug/24ug; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Changes in IL-6 Levels
Description: Changes in IL-6 Levels in the sputum supernatant compared to screening visit
Time Frame: Screening visit and 2 hours post inhalation of treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Formoterol (FORM) Total Dose 24ug: 2 puffs of Formoterol (FORM) 12ug (total dose 24ug)
- Symbicort® Total Dose 400ug/12ug: 2 puffs of a combination of formoterol (6ug) and ICS (Budesonide, (BUD) 200ug)
- Symbicort® Total Dose 800ug/24ug: 2 puffs of a combination of Formoterol (12ug) and budesonide (400ug)
- Pulmicort 800: 2 puffs of budesonide 400ug (total dose 800ug)
Arm/Group | Formoterol (FORM) Total Dose 24ug | Symbicort® Total Dose 400ug/12ug | Symbicort® Total Dose 800ug/24ug | Pulmicort 800
Number analyzed (Participants) | 13 | 13 | 13 | 12
pg/mL | -29 (25) | -14 (19) | -28 (22) | -29 (22)

3. Secondary Outcome: Changes in CXCL8 Levels
Description: Changes in CXCL8 concentrations in sputum compared to screening visit.
Time Frame: Screening visit and 2 hours post inhalation of treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Pulmicort 800: budesonide total dose 800ug
Arm/Group | Formoterol (FORM) Total Dose 24ug | Symbicort® Total Dose 400ug/12ug | Symbicort® Total Dose 800ug/24ug | Pulmicort 800
Number analyzed (Participants) | 13 | 12 | 12 | 12
ng/mL | -0.04 (0.35) | -2.1 (0.7) | -2.2 (0.55) | -1.5 (0.4)

4. Secondary Outcome: Changes in TNF Alpha
Description: Sputum TNF-alpha levels obtained from induced sputum compared to screening visit.
Time Frame: Screening visit and 2 hours post inhalation of treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Symbicort® Total Dose 800ug/24ug: 2 puffs of a combination of formoterol (12ug) and BUD (400ug)
- Pulmicort 800ug: budesonide total dose 800ug
Arm/Group | Formoterol (FORM) Total Dose 24ug | Symbicort® Total Dose 400ug/12ug | Symbicort® Total Dose 800ug/24ug | Pulmicort 800ug
Number analyzed (Participants) | 13 | 13 | 12 | 13
pg/mL | -4.8 (9.0) | -5.7 (7.9) | -7.8 (7.3) | -9.4 (7.4)

5. Secondary Outcome: Changes in Lung Function Parameter FEV1
Description: Improvement in FEV1 compared to baseline levels.
Time Frame: Baseline and 2 hours post inhalation
Measure: Mean (Standard Error); unit: mL
Groups:
- Symbicort® Total Dose 800ug/24ug:: 2 puffs of a combination of formoterol (12ug) and BUD (400ug)
Arm/Group | Formoterol (FORM) Total Dose 24ug | Symbicort® Total Dose 400ug/12ug | Symbicort® Total Dose 800ug/24ug: | Pulmicort 800ug
Number analyzed (Participants) | 30 | 30 | 30 | 30
mL | 160 (28) | 120 (25) | 200 (30) | 52 (18)

ADVERSE EVENTS:
Time Frame: 4 months
Description: All Adverse Events during the clinical investigation will be recorded and documented in the relevant section of the Case Report Form
Groups:
- Formoterol 24ug: Formoterol (FORM) total dose 24ug:
- Symbicort® Total Dose 400ug/12ug:: Symbicort® total dose 400ug/12ug: 2 puffs of combination formoterol (12ug) and BUD (200ug)
- Symbicort® Total Dose 800ug/24ug: Symbicort® total dose 800ug/24ug: 2 puffs of a combination of formoterol (12ug) and BUD (400ug)
- Pulmicort 800ug: budesonide total dose 800ug:
Arm/Group | Formoterol 24ug | Symbicort® Total Dose 400ug/12ug: | Symbicort® Total Dose 800ug/24ug | Pulmicort 800ug
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No